CLINICAL TRIAL: NCT07116447
Title: Impact of Repeated Exposure to Alcohol Health Warning Messages in a Real-world Online Retail Setting: Protocol For a Randomised Controlled Trial in Systembolaget App
Brief Title: Impact of Alcohol Health Messages in a Real-world Online Retail Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: World Health Organization (Other)
Collaborators: Systembolaget (Unknown)
Responsible Party: Principal Investigator, Daša Kokole, Principal Investigator, World Health Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-03328-01
Record Dates: First submitted 2025-08-06; First posted 2025-08-11 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Behaviour Change; Knowledge; Risk Perception; Emotional Response; Message Perception; Intentions; Sales
Keywords: alcohol; health warning; online supermarket; point-of-sale

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention group will be exposed to textual health warning messages currently mandated for use in printed alcohol advertisements under the Swedish Alcohol Ordinance (1994:2046). Messages will rotate, with each user exposed to a single message per session. The following eight messages will be included:
  Alcohol is addictive. Alcohol can cause damage to nerves and the brain. Alcohol can cause damage to the liver and pancreas. Alcohol can cause cerebral haemorrhage and cancer. Half of drivers who die in road traffic accidents involving just one vehicle are under the influence of alcohol.
  Half of all people who drown have alcohol in their blood. Alcohol consumption during pregnancy can damage the child. Children who are given alcohol at home drink to intoxication more frequently than other children.
  Interventions: Behavioral: Health messages - existing Swedish legislation
- Control (Active Comparator): The control group will consistently be exposed to health messages that are commonly present on existing alcohol labels and are aligned with voluntary commitments of alcohol producers, such as pictograms indicating no alcohol use during pregnancy and while driving. These pictograms will be displayed in black and white and in small sizes consistent with current practice, with a diameter of approximately 6 millimetres.
  Interventions: Behavioral: Health messages - pictograms

INTERVENTIONS:
Behavioral: Health messages - existing Swedish legislation — Textual health warning messages currently mandated for use in printed alcohol advertisements under the Swedish Alcohol Ordinance, focusing on communicated various alcohol harms
  Arms: Intervention
Behavioral: Health messages - pictograms — Pictograms indicating no alcohol use during pregnancy and while driving
  Arms: Control

SUMMARY:
The goal of this between-participants parallel randomized controlled trial conducted in the Systembolaget mobile application is to investigate the impact of exposure to health messages on cognition and behaviour.

The primary study objective is to examine whether repeated exposure to rotating health warning messages in a mobile app where customers can purchase alcoholic beverages influences the number of purchased units of alcohol over the studied period.

The secondary objectives are to examine whether repeated exposure to health warning messages in a mobile app influences the number of alcoholic and non-alcoholic products purchased over the studied period, knowledge of alcohol-related harms, alcohol-related risk perceptions, emotional response to the message, engagement with the messages, behavioural intentions and self-reported behaviour of the study participants.

Users of the app providing informed consent for participation in the study will be assigned either to an experimental group, where they will be exposed to rotating messages describing health risks associated with alcohol designed in line with the existing Swedish regulation, or to a control group that will be exposed to messages reflecting existing industry practice.

The intervention will last for ten weeks, during which the recruited participants' data on product purchases in the app will be collected through in-app analytics. Both the number of alcoholic units and number of products purchased per session will be assessed and compared at the session level between the two groups. At the end of the intervention, participants will complete a short survey examining their knowledge, risk perceptions, emotional response, engagement with the messages, intentions and behaviour.

ELIGIBILITY:
Inclusion Criteria:

* minimum alcohol purchase age in Sweden (20+)
* have downloaded the Systembolaget app and have given permission to the app to track in-app analytics
* understand Swedish language

Exclusion Criteria:

* not of minimum alcohol purchase age in Sweden
* no permission to track in-app analytics
* no understanding of Swedish language

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11719 (Actual)
Dates: Start 2025-09-02 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
Number of purchased units of alcohol | From enrolment to the end of the intervention period at 10 weeks
  Alcohol units will be calculated based on product-specific information on alcohol by volume (ABV) and volume purchased. The calculations will be made for the overall purchases and separately by type of beverage (beer, wine, spirits, other).

SECONDARY OUTCOMES:
Number of individual purchased products | From enrolment to the end of the intervention period at 10 weeks.
  For overall purchases and separately by type of beverage (beer, wine, spirits, other, non-alcoholic beverages)
Knowledge of alcohol-related harms | End of 10 week intervention period
  Will be assessed with question "Which of the following diseases and conditions does alcohol consumption increase the risk of? (select all that apply)", with the possible choices being [Cancer, Heart Disease , Liver Disease, Respiratory Disease, Alcohol use disorder, Injuries, Diabetes, Pancreatitis, Multiple sclerosis, Cerebral haemorrhage, Fetal alcohol spectrum disorder] displayed randomly, and "I don't know" and "None" as exclusive options. The question format and options were adapted from a previous study [18], but expanded with a longer list of possible outcomes described in the used health messages. Two outcomes will be derived from this question: (i) the correct identification of the conditions mentioned in the messages, with the possible score range being between 0 and 7 points, and (ii) the correct identification of cancer as condition that alcohol increases risk of.
Self-reported behaviour | End of 10 week intervention period
  Alcohol consumption behaviour will be based on question on whether they have foregone an alcoholic drink because they wanted to drink less and whether they have ever replaced alcoholic beverage with a non-alcoholic alternative because they wanted to drink less alcohol.
Risk perception | End of 10 week intervention period
  Perceived personal cancer risk will be measured with the question "If I consume alcohol on a regular basis, I am at greater risk of getting cancer." Perceived general health risk will be measured with the question "If I consume more alcohol, I am at greater risk for health harm". Both questions will be measured on 5-point Likert scale (Strongly Disagree to Strongly Agree).
Intention | End of 10 week intervention period
  Intention will be measured with the question "I intend to cut down on the number of alcohol units that I drink in the next month" on 5-point Likert scale (Strongly Disagree to Strongly Agree).
Emotional response | End of 10 week intervention period
  Emotional response will only be measured among those reporting to have noticed the warnings, "Thinking about messages I've seen as part of this study, I felt: disgusted / afraid / uncomfortable / worried / excited / pleased, with Likert answers scale from 1 to 5 (1 = Not at all, 3 = Moderately, and 5 = Very).
Engagement with messages | End of 10 week intervention period
  * Noticing, reading and recalling the warnings: Participants will be asked if they noticed health-related messages while using the Systembolaget app in the past two months. Participants will also be presented with a list of statements and asked to mark which of those have they been exposed to during participation in the study.
  * Information seeking behaviour: If participants noticed the health messages, they will be asked if they took any actions such as searching for more information about health risks, discussing the information with others, or looking for ways to reduce their alcohol consumption.
  * Message perceptions: Participants who noticed the health messages will also be asked to indicate their level of agreement with statements about the impact of the information on their alcohol consumption, purchasing behaviour, and their perception of the information's acceptability, novelty, relevance, and believability. Responses will be measured on a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Dasa Kokole, PhD, Principal Investigator — World Health Organisation Regional Office for Europe
Locations (1):
- Systembolaget mobile app, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in publications.
Supporting Information: Study Protocol, SAP
Time Frame: The dataset will be available following the open data sharing practices, and will be uploaded on Figshare repository (https://figshare.com/) once the article with the main results is published.
Access Criteria: Interested researchers will be able to access and download the data directly through the platform, without requiring any permissions. The article, including the dataset, will be shared under a noncommercial license (e.g. Creative Commons Attribution-NonCommercial (CC BY-NC)), allowing others to use the data for research, educational, or other noncommercial purposes, but not for commercial advantage or monetary gain.